CLINICAL TRIAL: NCT05419414
Title: The Use of Shear Wave Elastography, Transvaginal Ultrasound and Pelvic MRI in the Diagnosis of Adenomyosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Muhterem Melis Cantürk, Principal Investigator, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/1080
Record Dates: First submitted 2022-06-07; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Adenomyosis; Elastography; Transvaginal Ultrasound; Fibroid Uterus
MeSH Terms: conditions — Adenomyosis; Leiomyoma | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Adenomyosis (Active Comparator): Patients who were diagnosed with adenomyosis according to pelvic MRI were examined with transvaginal ultrasound. Certain ultrasonographic features of adenomyosis ( asymmetrical uterine wall thickening, myometrial cysts, fan shaped lines and shadows, presence of irregular junctional zone, presence of clue sign, global enlargement) were recorded. Then the patients were examined with shear wave elastography. Maximum and minimum median shear wave values were recorded through the selected regions of interest.
  Interventions: Device: Shear wave elastography
- Uterine Fibroid (Active Comparator): Patients who were diagnosed with myoma uteri according to pelvic MRI were examined with transvaginal ultrasound. Then the patients were examined with shear wave elastography. Maximum and minimum median shear wave values were recorded through the selected regions of interest.
  Interventions: Device: Shear wave elastography

INTERVENTIONS:
Device: Shear wave elastography — Both groups were examined with shear wave elastography.
  Other Names: elastography

SUMMARY:
In this prospective cohort study, the patients who were diagnosed with either uterine fibroid (control group) or adenomyosis (study group), were examined with transvaginal ultrasound and shear wave elastography. Definitive diagnosis was established by pelvic MRI. Shear wave elastography data of both groups were compared. Features of adenomyosis on transvaginal ultrasound were also recorded for study group.

DETAILED DESCRIPTION:
In this prospective cohort study, the patients who applied to the Gynecology and Infertility Outpatient Clinic in Istanbul University Faculty of Medicine between October 2018 and October 2021 due to abnormal uterine bleeding, pelvic pain, infertility were evaluated. The patients who were diagnosed with adenomyosis and uterine myoma according to clinical evaluation were included and grouped. Clinical diagnosis were confirmed with contrast enhanced pelvic magnetic resonance imaging. No histopathological confirmation were included in this study. 34 patients were included in adenomyosis group and 31 patients were included in myoma group. All patients were evaluated with shear wave elastography; 3 regions of interest were selected for each elastographic evaluation. Average shear values were determined automatically; then, minimum and maximum mean shear values were recorded accordingly. Elastography values of both groups were compared in order to detect any statistically significant difference between 2 groups. In addition to elastography evaluation, the compatibility of transvaginal ultrasound and magnetic resonance were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who applied to outpatient clinic due to abnormal uterine bleeding, pelvic pain, infertility.

Exclusion Criteria:

* Patients who are currently pregnant or has current malignancy, use combined oral contraceptives, gonadotropin releasing hormone agonist, intrauterine device or currently taking hormonal replacement therapy.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Both pathologies belong to female reproductive system.
Enrollment: 65 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Elastography data of adenomyotic lesions and fibroids | First we visualize the lesion in B-Mode ultrasound, then with the help of shear wave elastography, a color map is formed over the pathological lesion. We select 3 regions of interest to measure tissue stiffness. This takes about 15 minutes.
  By using shear wave elastography, we can calculate the stiffness of selected region of uterine pathology. We use transvaginal ultrasound probe while performing shear wave elastography. The selected region of interest is defined as 10 mm circular area which is selected by the ultrasonographer. Stiffness of the tissue is calculated by elastography program which works by emitting acoustic radiofrequency impulses. These impulses creates transversely oriented shear waves which propagates through the tissue. The velocity of the shear waves is measured by the device and by using Young's modulus, shear wave elastography provides us a numerical value in kiloPascal. This value gives us important information regarding the stiffness of the tissue. For adenomyotic lesions and fibroids, shear wave elastography is performed and for each selected region of interest, a numerical value in kilopascal is given by the ultrasound and we aim to compare these data for adenomyosis and fibroid groups

SECONDARY OUTCOMES:
Ultrasonographic features of adenomyotic lesions | This part consists of transvaginal ultrasound examination in B-Mode. This examination takes up to 20 minutes.
  To describe the features of adenomyosis seen during the transvaginal ultrasound examination, we perform a pelvic ultrasound using transvaginal probe in B-Mode. During the examination we analyze and record for the presence of certain features such asymmetrical uterine wall thickening, myometrial cysts, hyper echoic islands, fan-shaped shadowing, subendometrial buds and lines and irregular or interrupted junctional zone. We recorded presence and absence of each feature for every patient in adenomyosis group. At the end we we calculated the percentage of each feature's presence in patients diagnosed with adenomyosis. We listed the most common and least seen feature. We also recorded the presence of endometrioma or deep infiltrating endometriosis in order to calculate the percentage of patients in which adenomyosis and endometriosis coexist.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu X, Ding D, Ren Y, Guo SW. Transvaginal Elastosonography as an Imaging Technique for Diagnosing Adenomyosis. Reprod Sci. 2018 Apr;25(4):498-514. doi: 10.1177/1933719117750752. Epub 2018 Jan 10. PMID 29320956
- [Background] Stoelinga B, Hehenkamp WJ, Brolmann HA, Huirne JA. Real-time elastography for assessment of uterine disorders. Ultrasound Obstet Gynecol. 2014 Feb;43(2):218-26. doi: 10.1002/uog.12519. Epub 2014 Jan 12. PMID 23703939
- [Background] Vercellini P, Vigano P, Somigliana E, Daguati R, Abbiati A, Fedele L. Adenomyosis: epidemiological factors. Best Pract Res Clin Obstet Gynaecol. 2006 Aug;20(4):465-77. doi: 10.1016/j.bpobgyn.2006.01.017. Epub 2006 Mar 24. PMID 16563868
- [Background] Zhang Q, Duan J, Liu X, Guo SW. Platelets drive smooth muscle metaplasia and fibrogenesis in endometriosis through epithelial-mesenchymal transition and fibroblast-to-myofibroblast transdifferentiation. Mol Cell Endocrinol. 2016 Jun 15;428:1-16. doi: 10.1016/j.mce.2016.03.015. Epub 2016 Mar 15. PMID 26992563
- [Background] Ami O, Lamazou F, Mabille M, Levaillant JM, Deffieux X, Frydman R, Musset D. Real-time transvaginal elastosonography of uterine fibroids. Ultrasound Obstet Gynecol. 2009 Oct;34(4):486-8. doi: 10.1002/uog.7358. No abstract available. PMID 19790094
- [Background] Sarvazyan A, Hall TJ, Urban MW, Fatemi M, Aglyamov SR, Garra BS. AN OVERVIEW OF ELASTOGRAPHY - AN EMERGING BRANCH OF MEDICAL IMAGING. Curr Med Imaging Rev. 2011 Nov;7(4):255-282. doi: 10.2174/157340511798038684. PMID 22308105
- [Background] Gorgulu FF, Okcu NT. Which imaging method is better for the differentiation of adenomyosis and uterine fibroids? J Gynecol Obstet Hum Reprod. 2021 May;50(5):102002. doi: 10.1016/j.jogoh.2020.102002. Epub 2020 Nov 23. PMID 33242677
- [Background] Stoelinga B, Hehenkamp WJK, Nieuwenhuis LL, Conijn MMA, van Waesberghe JHTM, Brolmann HAM, Huirne JAF. Accuracy and Reproducibility of Sonoelastography for the Assessment of Fibroids and Adenomyosis, with Magnetic Resonance Imaging as Reference Standard. Ultrasound Med Biol. 2018 Aug;44(8):1654-1663. doi: 10.1016/j.ultrasmedbio.2018.03.027. Epub 2018 May 18. PMID 29784438
- [Background] Shwayder J, Sakhel K. Imaging for uterine myomas and adenomyosis. J Minim Invasive Gynecol. 2014 May-Jun;21(3):362-76. doi: 10.1016/j.jmig.2013.11.011. Epub 2013 Dec 4. PMID 24316138
- [Background] Leone FP, Timmerman D, Bourne T, Valentin L, Epstein E, Goldstein SR, Marret H, Parsons AK, Gull B, Istre O, Sepulveda W, Ferrazzi E, Van den Bosch T. Terms, definitions and measurements to describe the sonographic features of the endometrium and intrauterine lesions: a consensus opinion from the International Endometrial Tumor Analysis (IETA) group. Ultrasound Obstet Gynecol. 2010 Jan;35(1):103-12. doi: 10.1002/uog.7487. PMID 20014360
- [Background] Van den Bosch T, Dueholm M, Leone FP, Valentin L, Rasmussen CK, Votino A, Van Schoubroeck D, Landolfo C, Installe AJ, Guerriero S, Exacoustos C, Gordts S, Benacerraf B, D'Hooghe T, De Moor B, Brolmann H, Goldstein S, Epstein E, Bourne T, Timmerman D. Terms, definitions and measurements to describe sonographic features of myometrium and uterine masses: a consensus opinion from the Morphological Uterus Sonographic Assessment (MUSA) group. Ultrasound Obstet Gynecol. 2015 Sep;46(3):284-98. doi: 10.1002/uog.14806. Epub 2015 Aug 10. PMID 25652685
- [Background] Acar S, Millar E, Mitkova M, Mitkov V. Value of ultrasound shear wave elastography in the diagnosis of adenomyosis. Ultrasound. 2016 Nov;24(4):205-213. doi: 10.1177/1742271X16673677. Epub 2016 Oct 12. PMID 27847535

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT05419414/Prot_SAP_000.pdf